CLINICAL TRIAL: NCT06904352
Title: Reliability and Validity of Physical Tests and Musculoskeletal Ultrasound As an Add-on in Classifying Anterior Knee Pain
Acronym: AKP
Status: Not yet recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Joannes M Hallegraeff, Dr. in clinical epidemiology, Vrije Universiteit Brussel
Other Study IDs: 24361 AKP; Vrije Universiteit Brussel (Other: Vrije Universiteit Brussel)
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: musculoskeletal ultrasound-physical tests-anterior knee pain-reliability
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients with on-traumatic anterior knee pain in primary care physiotherapy and general practice: No interventions will be applied

SUMMARY:
Musculoskeletal ultrasound (MSU) or sonography is a non-invasive diagnostic technique and can extend the clinical examination of Anterior Knee Pain by visualizing musculoskeletal pathology to detect invisible flaws, it is safe, cheap and easy to use in primary care and therefore ensuring substitution of care. The European Society of Musculoskeletal Radiology (ESSR) has concluded that MSU can accurately classify APK pathologies. Protocol-based MSU can detect pathologic changes including cartilage swelling, fragmentation of the tibial tubercle ossification center, patellar tendon lesions, and reactive bursitis of the deep or superficial tibial patellar bursae and is increasingly used by physical therapists in the diagnostic process.

It is hypothesized that the validity of the physical examination is insufficient to accurately classify different conditions in AKP in patients aged 7-50 years. Therefore the use of MSU as an add-on is essential.

The purpose of this study is at first to assess the validity of the physical examination and second to evaluate the inter-rater reliability of protocol-based MSU and physical examination, in patients with AKP, in primary care physiotherapy.

The study is a cross-sectional observational study with four measurements within 60 minutes, without any intervention, performed with a single-gate diagnostic design with the same eligibility criteria for all participants including one group for comparison and measurement. The Strengthening the Reporting of Observational Studies in Epidemiology Statement was used as a guideline.

DETAILED DESCRIPTION:
Data will be collected from April 2025 to November 2025 in two multidisciplinary healthcare centers in the Netherlands, Amsterdam and Amersfoort. All confidential records were stored in a secure area with access only to JMH and HvdP, who also prepared the database for data analysis, to guarantee anonymity and confidential input of all data. In all participants, the sequence of measurements was identical. Pseudo anonymization was done by using the initials of the examiners and inclusion number.

Confidentiality and anonymity were guaranteed by storing all records in a secure area, and an encrypted electronic database was used for all encoded data. Patient Reported Outcomes Measures (PROMs) and physical tests are to be administered during the same time of day. They followed a predetermined order as outlined on the data registration form.

ELIGIBILITY:
Eligibility criteria are subjects, aged 7 to 50 years, with clinically confirmed non-traumatic anterior knee pain (AKP). Subjects must be able to read, understand, and speak Dutch. Before participation, the study protocol was expressed verbally and in writing, and subsequently informed consent was obtained. In addition, we assessed whether participants did understand it.

Inclusion Criteria:

* All consecutive patients presenting clinical symptoms of AKP were screened for eligibility.

Exclusion Criteria:

* patients with knee effusion, patients having patella instability, surgeries or previous fractured knee joint in the past, systemic pathology including inflammatory joint disease, and patients with interventions in the last three months including corticosteroid injection or physiotherapy.

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants in primary care with non-traumatic anterior knee pain
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Reliability and validity of physical tests and musculoskeletal ultrasound as an add-on in classifying anterior knee pain | From April 2025 to October 2025 or until the end of the study
  Measurements are taken in primary care in the Netherlands in two different healthcare settings and are taken in two ways: at first physical tests and at second using musculoskeletal ultrasound to diagnose patients with anterior knee pain.

CONTACTS AND LOCATIONS:
Overall Officials: Joannes M Hallegraeff, MSc, PhD, Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided
This is an initial study who focus on this topic. We first want to assess whether the data is adeqauate enough to possibly share with other researchers. We are not thinking of doing so for the time being.